CLINICAL TRIAL: NCT04346043
Title: Strain Study: To Access the Egyptian COVID-19 Whole Genome (Dominant Strain) by Next Generation Sequencing (NGS) and Compare to the International Worldwide Database
Brief Title: To Access the Egyptian COVID-19 Whole Genome by NGS and Compare to the International Worldwide Database
Acronym: Strain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hesham Elghazaly,MD, Director of Faculty of Medicine Ain Shams University Research Institute, Ain Shams University
Other Study IDs: FMASU P16a/ 2020
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Coronavirus Disease (COVID-19)
Keywords: Egypt
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Nasopharyngeal & oropharyngeal swabs will be taken from patients with COVID-19
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an exploratory study that will be performed on confirmed positive COVID-19 samples to identify the dominant viral genome strain in Egyptians using next generation sequencing (NGS).

DETAILED DESCRIPTION:
CASE SELECTION:

100 cases of COVID-19 samples proved to be positive in Ain Shams University Specialized Hospital labs (at the Universities reference lab) will be tested in the strain study.

Detection of virus:

Sample collection:

Nasopharyngeal & oropharyngeal swabs will be taken from suspected cases and put in a specific viral transpot media.

One oropharyngeal swab (OS) and one nasopharyngeal swab (NS) are collected from hospitalized SARI patients (adults and pediatric) and then added together in one 15ml Falcon tube containing 2ml viral transport media (VTM). The swabs are obtained by a well-trained doctor or medical professional.

Oropharyngeal swabbing: A dry sterile tip flocked with nylon fiber swab applicator is used to swab both the tonsils and the posterior pharynx. The swab is placed in a 15 ML Falcon tube labeled with the patient unique ID and containing 2ml VTM (consisting of sterile solution of bovine albumin fraction V, HEPES buffer, penicillin and streptomycin in HANK's balanced salt solution). The applicator stick is then cut off.

Nasopharyngeal swabbing: A flexible, sterile tip flocked with nylon fiber swab applicator is inserted into the nostril and back to the nasopharynx and left in place for a few seconds. It is then slowly withdrawn with a rotating motion. The swab is inserted in the same tube as the throat swab and the shaft is cut.

Sample procedures:

The tube containing the nasopharyngeal and oropharyngeal swab will be agitated vigorously for 10 seconds using a vortex mixer. Both swabs should then be removed from the tube and discarded using sterile forceps that should be sterilized from one sample to another to avoid cross contamination.

The resulting supernatant (VTM/UTM) is decanted in 2 cryogenic vials labeled with the patient ID.

One cryogenic vial will be immediately stored at -70°C freezer or lower temperature such as liquid nitrogen tank for QA and further characterization of the COVID-19.

The other vial will be tested according to the lab capacity:

VIRAL RNA ISOLATION:

Using commercially available kits supplied by thermofisher or other recommended companies. Work will be done in Biosafety level 2 cabinets under complete sterile conditions.

COVID-19 DETECTION:

Using real time reverse transcription polymerase chain reaction (rRT-PCR) the test can be done on respiratory samples obtained by various methods, including nasopharyngeal swab or sputum sample. Results are generally available within a few hours. Molecular methods leverage polymerase chain reaction (PCR) along with nucleic acid tests, and other advanced analytical techniques, to detect the genetic material of the virus using real-time reverse transcription polymerase chain reaction for diagnostic purposes. Commercially available kits supplied by HVD, thermofisher and others.

Coronavirus Research Using Next-Generation Sequencing (NGS) One assay surveying the entire coronavirus genome for epidemiological investigation: A major challenge for microbiologists and virologists is the prediction of patterns of evolution and emergence of disease agents. RNA viruses like the coronavirus share the biological feature of high genetic variability, which causes them to appear as clouds of mutants. Coronavirus variants also emerge through antigenic shift within animal reservoirs, such as bats and snakes. Ion Torrent targeted next-generation sequencing (NGS) enables a streamlined research workflow for complete genome sequencing and epidemiological studies of SARS-CoV-2 (the coronavirus responsible for COVID-19). Through the use of a set of highly specific, universal coronavirus primers in combination with a high-fidelity master mix, all genomic segments are amplified and the DNA amplicons are sequenced on any Ion Torrent system to deliver highly accurate coronavirus typing in under a day.

The Ion AmpliSeq SARS-CoV-2 Research Panel consists of 2 pools with amplicons ranging from 125-275 bp in length for complete viral genome sequencing and variant detection.

Bioinformatic analysis of the NGS DATA Next-generation sequencing, or NGS, can generate enormous amounts of data, and the challenge becomes finding ways to analyze it properly. In this study we are going to use some bioinformatic tools to analyze and track the outbreak in Egypt.

Genome Detective bioinformatic tool, Takes the raw data from the sequencing machine, filter out results from non-viruses, piece together the genome and use that to identify the virus. It does not rely on any prior guesses or hypotheses, so it can even identify viruses that have not been seen before. This was used to confirm the first case of COVID-19 in Belgium, identifying it as a SARS-related coronavirus.

NextStrain, is an online resource that uses genome data to monitor the evolution of disease-causing organisms such as viruses in real time. It has tracked several outbreaks including Zika, Ebola and Dengue and has even been used to inform World Health Organization policy on seasonal flu.

NextStrain already has over 700 genomes of the new coronavirus, which it can use to trace the outbreak by detecting new mutations in the virus. The mutations do not necessarily affect how the virus behaves, but they can act as a genetic signature to link cases that are related. Like tracing your ancestry through a DNA test, a virus sequenced in Madrid, for instance, could have mutations that suggest it originated from an outbreak in Italy.

Sequencing cases will become even more important because as we start cracking down on (the pandemic), which we hopefully will achieve, it will tell us how many transmission chains are still circulating and whether the virus is being transported from one region to another.

Phylogenetic analysis of these 2019-nCoV genomes and those of other coronaviruses to be completed by virology consultant

Multiple sequence alignment will be performed with the ClustalW program using MEGA software (version 7.0.14). Phylogenetic trees will be constructed by means of the maximum-likelihood method with MEGA software (version 7.0.14). The full-genome viral sequences will be deposited in the dataset of Global Initiative on Sharing All Influenza Data (GISAISD, No. EPI_ISL_402123, EPI_ISL_403928-31).

ELIGIBILITY:
Inclusion Criteria:

Patients With confirmed COVID-19

Exclusion Criteria:

inadequate sample of the patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 cases of COVID-19 samples proved to be positive in Ain Shams University Specialized Hospital labs (at the Universities reference lab) will be tested in the strain study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-20 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Dominant viral genome strain | 9 months
  Identify the dominant viral genome strain in Egyptians With COVID-19 infection using next generation sequencing (NGS)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ain Shams University Research Institute- Clinical Research Center, Cairo, Non-US, Egypt

IPD SHARING:
Plan to Share IPD: No